CLINICAL TRIAL: NCT06729203
Title: Effect of Ultrasound Cavitation on Insulin Resistance in Patients with Central Obesity in Female
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aya Saeed Khalil Shazly, physiotherapist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 012/005421
Record Dates: First submitted 2024-12-08; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Central Obesity
Keywords: central obesity; ultrasound cavitation; insulin resistance; HOMA ir
MeSH Terms: conditions — Obesity, Abdominal; Insulin Resistance | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): this group receive ultrasound cavitation on abdominal muscles
  Interventions: Device: Ultrasound cavitation
- Group B (Active Comparator): received aerobic exercises and low caloric diet treatment.
  Interventions: Other: Exercise

INTERVENTIONS:
Device: Ultrasound cavitation — Ultrasound Fat Cavitation (USFC) is the method in handling obesity, especially in destroying fat and shaping a particular part of the body. As one of the non-surgical correction methods, USFC is preferred at decreasing the risk of complications due to obesity.
  Other Names: Ultrasound Fat Cavitation (USFC)
  Arms: Group A
Other: Exercise — The female will stand on the cushioned tread and grasp by her both hands the two arms of the treadmill. Treadmill will adjust to apply moderate intensity training. It was used for 30 minutes divided into five-minutes warming up, twenty-minutes active exercise and five-minutes cooling down and it was used twice a week for twelve weeks.
  Other Names: aerobic exercise
  Arms: Group B

SUMMARY:
The purpose of this study was to investigate the effect of ultrasound cavitation on insulin resistance, HbA1c and skin fold in patients with abdominal central obesity.

DETAILED DESCRIPTION:
Few researchers have detected the effects of ultrasonic cavitation on insulin resistance in subjects with central obesity. However, there were many conflicts and no clear evidence in the literature concerning the superiority of cavitation on body contour adjustment. Consequently, this study aimed to investigate the effects of ultrasound cavitation, aerobic exercise and a low-calorie dietary program on insulin resistance and total plasma HOMA ir and body contouring in female with abdominal obesity.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects with central obesity.
* Female participants aged between 25 to 40 years.
* Body Mass Index (BMI) ranged from 30 to 35 kg/m2 as high BMI indicates more obesity and central obesity.
* Waist circumference greater than 88 cm, indicative of abdominal obesity.
* Diagnosed with insulin resistance (HOMA-IR > 2.9).
* Sedentary lifestyle, defined as engaging in less than 150 minutes of moderate-intensity physical activity per week.
* Willingness to provide informed consent and comply with study procedures.

Exclusion Criteria:

* • Subjects diagnosed with DM (HbA1c more than 6.5%).

  * History of metabolic disorders such as type 1 diabetes or thyroid disorders.
  * Subjects with BMI less than 30 kg/m2.
  * Subjects diagnosed with heart disease, liver as well as kidney diseases.
  * Subjects who take oral contraceptives.
  * Subjects with gestational Diabetes.
  * Pregnant or breastfeeding women were excluded from the study.
  * Use of weight-loss medications or supplements within the past six months.
  * Previous surgical procedures for weight loss or body contouring.
  * Contraindications to ultrasound therapy (e.g., metal implants in the abdomen, active skin infections).
  * Participation in another clinical trial within the last three months.

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
HOMA ir | "From enrollment to the end of treatment at 8 weeks"
  This study will evaluate changes in HOMA-IR from baseline to assess improvements in insulin sensitivity because of the ultrasound cavitation intervention.

SECONDARY OUTCOMES:
Skin fold by caliper | "From enrollment to the end of treatment at 8 weeks"
  The skinfold measurements will be taken using a Lange Skinfold Caliper, which provides accurate and reliable readings
Waist circumference (WC) by tape measurement | "From enrollment to the end of treatment at 8 weeks"
  Waist circumference (WC) is an essential anthropometric measure used to evaluate abdominal obesity. It serves as an indicator of visceral fat, which is associated with a higher risk of metabolic disorders, including insulin resistance, type 2 diabetes, and cardiovascular diseases. By measuring waist circumference.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Giza, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided